CLINICAL TRIAL: NCT00518050
Title: Melanoma Survivors: Health Behaviors, Surveillance, Psychosocial Factors, and Family Concerns
Brief Title: Health Behaviors, Surveillance, Psychosocial Factors, and Family Concerns
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 06-128
Record Dates: First submitted 2007-08-15; First posted 2007-08-17 (Estimated); Last update posted 2015-07-16 (Estimated); Status verified 2015-07

CONDITIONS: Melanoma; Survivors; Psychological Factors
Keywords: Health Behaviors; Surveillance; 06-128
MeSH Terms: conditions — Melanoma; Health Behavior | interventions — Focus Groups; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- Specific Aim 1- Focus Group: Conduct focus groups in melanoma survivors to enhance the understanding of the behavioral aspects of:
  * Screening, skin self-examination, sun protection, and other cancer preventive practices;
  * Cognitive factors (knowledge, awareness, melanoma worry, and perceived risk) related to screening and sun protection practices; and,
  * Impact of melanoma on quality of life, family relationships, and economic issues arising from treatment
  Interventions: Behavioral: Focus group
- Specific Aim 2- Survey Study: A separate random sample of melanoma survivors will complete the pilot questionnaire. To enhance completion rates, survey instruments will be developed to be both self-administered and interviewer-administered. The survey will include questions from existing surveys, regarding demographics, sun sensitivity, eye and hair color, color of untanned skin, sun exposure, skin selfexamination, sun protection practices and frequency of sunburns, psychosocial/cognitive factors: skin cancer knowledge, skin awareness, cancer worry, perceived risk of recurrence, cancer risk and screening behaviors, and access to health care and insurance.
  Interventions: Behavioral: Survey

INTERVENTIONS:
Behavioral: Focus group — Conduct focus groups in melanoma survivors to enhance the understanding of the behavioral aspects of:
  * Screening, skin self-examination, sun protection, and other cancer preventive practices;
  * Cognitive factors (knowledge, awareness, melanoma worry, and perceived risk) related to screening and sun protection practices; and,
  * Impact of melanoma on quality of life, family relationships, and economic issues arising from treatment
  Groups: Specific Aim 1- Focus Group
Behavioral: Survey — History of sun exposure Medical factors Affect, cognition, and quality of life Behavioral adoption Demographics Phenotypic factors Economic/healthcare factors
  Groups: Specific Aim 2- Survey Study

SUMMARY:
The purpose of this study is to examine the health behaviors of melanoma survivors. We want to know about their thoughts and concerns. Melanoma is a type of skin cancer. The number of people being diagnosed with melanoma is growing. Many people who are diagnosed with melanoma are young. Little research has been done to find out how melanoma survivors feel years after they have been treated.

DETAILED DESCRIPTION:
The rapidly rising incidence and mortality rates of melanoma, the most fatal form of skin cancer, are among the greatest increases of all preventable cancers over the past decade. However, because of recent advances in early detection, secondary prevention efforts, and treatment, the number of melanoma survivors is increasing. Little research has been conducted on melanoma survivors and important opportunities exist for research in this understudied population. Understanding recurrence and second primary cancer risk, cognitive characteristics, behaviors, surveillance patterns, economic sequelae, and family issues of melanoma survivors is imperative from a public health standpoint to promote the health and well-being of this cohort. The objectives of this study are to: 1) conduct focus groups to enhance our understanding of the behaviors of melanoma survivors, and 2) conduct a pilot survey study based on the results of the focus groups to further describe the behavioral and psychosocial issues in melanoma survivors. This will be among the first studies that explores behavioral and psychosocial issues in melanoma survivors. The study findings will inform a large-scale melanoma survivorship grant proposal to the National Cancer Institute or other federal/private sources of funding.

ELIGIBILITY:
Inclusion Criteria:

For the focus group recruitment (Specific Aim 1) - Patients with melanoma (invasive primary cutaneous melanoma, stages 1-III), who have been treated at MSKCC from 1996-2005

For the survey group recruitment (Specific Aim 2):

patients with melanoma (invasive primary cutaneous melanoma, stages 1-III), who have been treated at MSKCC from 2001-2011• Ability to sign informed consent which indicates the psychosocial, behavioral, epidemiological nature of this study

• Age ≥ or = to 18 years and fluent in the English language

Exclusion Criteria:

* Patients with intraepithelial (in situ) melanoma

  * Patients with stage IV melanoma
  * Patients with nodal or visceral melanoma without a documented primary lesion
  * Patients with prior malignancies For the focus group recruitment (Specific Aim 1): (patients treated at MSKCC from 1996-2005) who have a diagnosis >10 years ago from treatment. For the survey group recruitment (Specific Aim 2): patients treated at MSKCC from 2001-2011)who have a diagnosis >10 years ago from treatment.
  * Patients with a recent diagnosis of melanoma, <12 months
  * Patients who are one year or more post diagnosis and are still receiving treatment for their melanoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible melanoma survivors will be initially identified and screened using the Melanoma DMT Database. We will select a random sample from the database.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2006-10; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
This pilot study will provide baseline data to enhance our understanding of the behaviors of melanoma survivors. | 2 hours

SECONDARY OUTCOMES:
Conduct a pilot survey study of melanoma survivors to describe the behavioral and psychosocial issues in melanoma survivors. Results from the survey will enable us to obtain preliminary data in order to conduct a larger scale study. | half an hour

CONTACTS AND LOCATIONS:
Overall Officials: Susan Oliveria, ScD, MPH, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center 1275 York Avenue, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org